CLINICAL TRIAL: NCT03881189
Title: Efficacy and Tolerance Evaluation of an Intradermal Injective Treatment for the Area Around the Eyes
Brief Title: Efficacy and Tolerance Evaluation of an Injective Treatment for the Area Around the Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Principal Investigator, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1518
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Under-eyes Dark Circles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUNEKOS ® 200 (Experimental): The 1st intradermal treatment (T1i) with "Sunekos ® 200" was carried out during the basal visit (T0), after basal evaluations planned by the study procedure, and then repeated 2 more times with an interval of 15 days (T2i and T3i)
  Interventions: Device: SUNEKOS® 200

INTERVENTIONS:
Device: SUNEKOS® 200 — The intradermal injection procedure was performed bilaterally, on the area around the eyes including the eyelids, using periosteal and subepidermal injection techniques. This injective procedure consists of micro-wheals of 0.2 ml just above the periosteum and micro-wheals of 0.1 ml very superficially, just under epidermis.

SUMMARY:
Efficacy and tolerance evaluation of an intradermal injective HA and aminoacids based treatment for the area around the eyes

DETAILED DESCRIPTION:
Primary end point of this study was to evaluate clinically and by non-invasive instrumental measurements the aesthetic performance on the area around the eyes of the"SUNEKOS® 200" injective treatment. Precisely three micro-injection sessions with an interval of 15 days were performed by a specialized dermatologist using periosteal and subepidermal injection techniques, on the area around the eyes of female volunteers with dark circles.

An additional aim of this study is to evaluate the product tolerance by both the investigator and volunteers.

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* 30-65 years,
* dark circles,
* available and able to return to the study site for the post-procedural follow-up examinations;
* agreeing to present at each study visit without make-up;
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products;
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the informed consent form

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol or drug abusers;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test at T0 (before the 1st aesthetic procedure) and at T3i (1 month after the 1st injection treatment execution, before the 3rd aesthetic procedure);
* Body Mass Index (BMI) variation (± 1) during the study period;
* performing skin treatments for aesthetic correction (biomaterials implants, face lifting, botox injections, laser, chemical peeling) in the 6 months prior to the study start;
* performing permanent filler in the past;
* change in the normal habits regarding food, physical activity, face cosmetic, cleansing and make-up use during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 9 months.
* Dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne).
* Diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy.
* Anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of wrinkles grade around the eyes | T0 (baseline), T3i+1 (1 day after the 3rd injection treatment with Sunekos 200), T2M (after 2 months), T3M (after 3 months)
  Visual score of crow's feet, according to a reference photographic scale from 0 (no wrinkles) to 7 (very marked wrinkles)
Change from baseline of dark circles grade | T0 (baseline), T3i+1 (1 day after the 3rd injection treatment with Sunekos 200), T2M (after 2 months), T3M (after 3 months)
  Visual score of dark circles grade, according to a reference photographic scale from 0 (absent) to 4 (very marked)
Change from baseline of roughness profilometric parameters | T0 (baseline), T3i+1 (1 day after the 3rd injection treatment with Sunekos 200), T2M (after 2 months), T3M (after 3 months)
  Crow's feet profilometric parameters measured by Primos compact portable device (GFMesstechnik). Ra is average roughness of the analysed profile, Rt is wrinkles total high, Rv is wrinkles maximum depth.
Change from baseline of dark circles colorimetric parameters | T0 (baseline), T3i+1 (1 day after the 3rd injection treatment with Sunekos 200), T2M (after 2 months), T3M (after 3 months)
  Dark circles colorimetric measured by Chroma Meter CR-200® . L* represent the lightness of the colour, a* represent the red component of the colour, b* represent the dark component of the colour
Change from baseline of spectrophotometrical value | T0 (baseline), T3i+1 (1 day after the 3rd injection treatment with Sunekos 200), T2M (after 2 months), T3M (after 3 months)
  Dark circles spectrophotometrical color value measured by a visible-UV-IR spectrophotometer

SECONDARY OUTCOMES:
change from of photographic documentation | T0 (baseline), T3i+1 (1 day after the 3rd injection treatment with Sunekos 200), T2M (after 2 months), T3M (after 3 months)
  Photographic documentation of the area around the eyes

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy